CLINICAL TRIAL: NCT07055906
Title: Developing and Testing a Video-feedback Intervention to Promote Racial-Ethnic Socialization Competency in Latino/a/x Families
Brief Title: Video-feedback Intervention to Promote Racial-Ethnic Socialization Competency (VIP-RACE)
Acronym: VIP-RACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Chardee Galan, Principal Investigator, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00025027; R21MD018693 (NIH)
Record Dates: First submitted 2025-06-11; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms; Anxiety Symptoms; Conduct Problems
Keywords: parenting program; Latino/a/x/é; racial-ethnic socialization
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video-feedback Intervention to Promote Racial-Ethnic Socialization CompEtency (VIP-RACE) (Experimental): All parent-child dyads will be assigned to the VIP-RACE parenting program.
  Interventions: Behavioral: Video-feedback Intervention to Promote Racial-Ethnic Socialization CompEtency (VIP-RACE)

INTERVENTIONS:
Behavioral: Video-feedback Intervention to Promote Racial-Ethnic Socialization CompEtency (VIP-RACE) — VIP-RACE is a brief, strengths-based, video-feedback intervention that targets parental racial-ethnic socialization (RES) motivation and competency in parents of 10-to-14-year-old Latino/a/x/e youth. Intervention sessions include: (1) Youth and parent assessment including videotaped parent-adolescent RES conversations; (2) Parent interview; and (3) Video feedback session during which parents and RES coaches review clips from the RES interaction tasks. Video feedback highlights parents' RES strengths and when sensitively applied, encourages parents to examine missed opportunities for engaging in RES. RES coaches emphasize that through the provision of cultural socialization and preparation for bias messages, parents can help protect their children from the damaging effects of discrimination and support positive racial-ethnic identity development. Parents develop a personalized action plan with goals and have the opportunity to receive up to 3-5 follow-up sessions to strengthen RES skill
  Other Names: Resiliencia y Apoyo hacia la Identidad Cultural, Educación y Superación juvenil (RAÍCES)

SUMMARY:
The aim of this study is to evaluate a novel cultural strengths parenting program - the Video-feedback Intervention to Promote Racial-Ethnic Socialization CompEtency (VIP-RACE) - which seeks to support Latine parents' motivation to engage in racial-ethnic socialization (RES) and strengthen their RES competency (improved skills and confidence, decreased stress). In the preliminary phases of this project, we iteratively refined the VIP-RACE program in partnership with advisory boards of youth, parents, and providers. The refined intervention will now be tested with five parents of 10-14-year-old Latine youth to identify gaps in the curriculum and obstacles to implementation that can be addressed prior to a larger pilot. The investigators will then conduct a proof-of-concept single-arm trial with Latine families to assess the feasibility, acceptability, and preliminary efficacy of VIP-RACE. The investigators hypothesize that VIP-RACE will be shown to be feasible and acceptable to families. The investigators also predict that bolstering parents' RES motivation and competency will result in increased frequency and quality of these conversations between parents and youth which, in turn, are expected to strengthen youth racial-ethnic identity and coping and have cascading effects on mental and behavioral health.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent is 10-to-14 years old (inclusive)
* Adolescent and parent are Latino/a/x/e or Hispanic
* Parent and youth have the capacity to provide consent/assent
* One parent is willing to participate
* Families must be willing to be video or audio recorded for the parent-child interaction task
* Youth and parent(s) must be willing to participate as dyads.
* Primary language of parent and adolescent is English and/or Spanish

Exclusion Criteria:

* Parent or adolescent has an intellectual disability, autism spectrum disorder, or other disorder that may limit ability to complete study (surveys and interviews require sustained attention, mental processing, and comprehension).
* Adolescent is not 10-to-14 years old
* Adolescent and/or parent are not Latino/a/x/e or Hispanic
* Primary language of parent and/or adolescent is not English and/or Spanish
* Youth and parent(s) are not willing to participate as dyads
* Family participated in Phase 1 of the study

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Quantitative) | Immediately after the intervention
  An adapted version of the Feasibility of Intervention Measure will obtain parents' feedback on the perceived feasibility of VIP-RACE. The Feasibility of Intervention Measure consists of five items scored on a 5-point Likert scale (e.g., "This program is easy to use") and demonstrates acceptable reliability. The measure will also include space for participants to provide open-ended feedback. The minimum value for this measure is 1 and the maximum value for this measure is 5, with higher scores indicating better outcomes.
Acceptability (Quantitative) | Immediately after the intervention
  An adapted version of the Acceptability of Intervention Measure will obtain parents' feedback on the perceived acceptability of VIP-RACE. The Acceptability of Intervention Measure consists of five items scored on a 5-point Likert scale (e.g., "I like this program") and demonstrates acceptable reliability. The measure will also include space for participants to provide open-ended feedback on which aspects of VIP-RACE were the most and least useful. The minimum value for this measure is 1 and the maximum value for this measure is 5, with higher scores indicating better outcomes.
Feasibility and Acceptability (Qualitative) | Immediately after the intervention
  A subgroup of parent participants (n=10-15) will complete semi-structured qualitative exit interviews to provide more in-depth feedback on their experience participating in the intervention. The interview will probe parents' views of the program, including what they found most and least useful, how the program helped them navigate RES conversations, barriers to participation, and suggestions for improving implementation in the future. The investigators will also include questions to explore variation in parents' RES practices, perceptions of program, and intervention impact based on youth and parent sex, and will also conduct semi-structured interviews with RES coaches to further assess feasibility and acceptability and guide refinements for a larger efficacy trial. The investigators will collect critical information that can be used in future trials, including barriers and facilitators to implementing the intervention and modifications that can be made to the program.
Feasibility (Attendance tracking) | Through study completion, an average of 9 weeks
  Participant attendance of VIP-RACE sessions will be tracked. VIP-RACE will be judged feasible if at least 75% of participants complete all three sessions of the program.
Change in Parental Racial-Ethnic Socialization (RES) Motivation | Baseline, immediately after the intervention, and 1-month follow-up
  An adapted version of the Motivation to Change Scale will assess parent-reported parental motivation to engage in RES with their children (e.g., "How important is it for you to talk to your child about discrimination they may experience"). The minimum value for this measure is 1 and the maximum value for this measure is 6, with higher scores indicating better outcomes.
Change in Parental RES Competency | Baseline, immediately after the intervention, and 1-month follow-up
  The Racial Socialization Competency Scale will assess parent-reported parental RES competency. The measure comprises 28 items (e.g., "teach my child to resolve a negative racial encounter with their peers."), and for each item, parents are asked to rate their confidence ("I believe I can"), skills ("I am/would be prepared to"), and stress ("I am/would be stressed to"). Parents respond using a 5-point Likert scale, with the lowest endorsement corresponding to the least confident, prepared, and stressed. Subscales include RES confidence, RES skill, and RES stress. The measure has been validated with diverse racial-ethnic groups, including with Latino/a/x caregivers (validation paper under review). The minimum value for this measure is 1 and the maximum value for this measure is 5, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Change in Parental RES Frequency | Baseline, 1-month follow-up
  The Ethnic-Racial Socialization Scale (minimum value 1, maximum value 5) and the Familial Ethnic Socialization Measure (minimum value 1, maximum value 5) will assess the frequency of parent- and youth-reported parental RES, specifically cultural socialization and preparation for bias messages. These measures have been adapted, validated, and utilized with diverse racial-ethnic groups since 1997 and 2001, respectively. Higher scores on both of these measures indicate better outcomes.
Change in Parental RES Quality | Baseline, 1-month follow-up
  The Observational Paradigm for Ethnic-Racial Socialization will be used to assess the quality of parents' cultural socialization and preparation for bias messaging. Specifically, parents and youth will be videotaped engaging in conversations about topics such as discrimination. Interactions will be coded using the Observational Measure for Ethnic-Racial Socialization, the companion coding system to the Observational Paradigm for Ethnic-Racial Socialization observational paradigm. The Observational Measure for Ethnic-Racial Socialization uses macro rating, a method that requires observers to synthesize interactions and apply a global impression on a 9-point scale (minimum value 1, maximum value 9). It includes codes for cultural socialization and preparation for bias (discrimination awareness and racial-ethnic coping strategies). Higher scores on this measure indicate better outcomes.
Change in Positive and Harsh Parenting during RES Conversations | Baseline, 1-month follow-up
  The investigators will assess global aspects of parenting (e.g., positive, harsh parenting) as observed during videotaped dyadic discussions of topics such as discrimination.
Change in Youth Racial-Ethnic Coping | Baseline, 1-month follow-up
  The Discrimination Coping Strategies Scale will assess parent- and youth-reported youth strategies for coping with racial-ethnic discrimination. The 6-item scale (minimum value = 1, maximum value = 5) includes two subscales, proactive coping and secondary coping, and has been validated for use with Latino/a/x youth. Higher scores on this measure indicate better outcomes.
Change in Youth Racial-Ethnic Identity | Baseline, 1-month follow-up
  The Ethnic Identity Scale will assess youth-reported youth racial-ethnic identity. The 17-item scale (minimum value = 1, maximum value = 4) includes three subscales, exploration, resolution, and affirmation, and has been validated for use with Latino/a/x youth. Higher scores on the exploration and resolution subscales indicate better outcomes, while lower scores on the affirmation susbscale indicates better outcomes.
Change in Youth Depressive and Anxiety Symptoms | Baseline, 1-month follow-up
  The Revised Child Anxiety and Depression Scale will assess parent- and youth- reported youth depressive and anxiety symptoms. The measure has been validated for use with children between 8 and 18 years of age. This measure has a minimum value of 0 and a maximum value of 2, with lower scores indicating better outcomes.
Change in Youth Conduct Problems | Baseline, 1-month follow-up
  The Strengths and Difficulties Questionnaire will assess parent- and youth- reported conduct problems. The Conduct Problems Scale will be used which includes items about rule-breaking and aggressive behaviors. The maximum value for this measure is 2 and the minimum value is 0, with lower scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — The Pennsylvania State University
Locations (1):
- Parents and Children Together (PACT) Lab Space, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual and aggregate survey data (including raw and recoded data) will be shared. The de-identification process will remove direct and indirect respondent identifiers. Once data are confirmed final, respondent identifiers will be deleted. Transcripts from interviews will be de-identified and sensitive content redacted where identification is plausible. These de-identified and redacted transcripts and coding summaries will be shared. Attendace data will also be shared.
  Following generation and quality check of raw transcripts from interviews, digital voice recordings will be permanently deleted to protect participant privacy. Respondent identifiers will not be shared. Raw transcripts and parent-child interaction task videos will be maintained but not shared. Transcripts from interviews and tasks will be de-identified and sensitive content redacted where identification is plausible. These de-identified and redacted transcripts and coding summaries will be shared.

REFERENCES:
- [Background] Kalofonos I, McCoy M, Altman L, Gelberg L, Hamilton AB, Gabrielian S. A Sanctioned Encampment as a Strategy for Increasing Homeless Veterans' Access to Housing and Healthcare During the COVID-19 Pandemic. J Gen Intern Med. 2023 Jul;38(Suppl 3):857-864. doi: 10.1007/s11606-023-08124-4. Epub 2023 Jun 20. PMID 37340271
- [Background] Vindrola-Padros C, Johnson GA. Rapid Techniques in Qualitative Research: A Critical Review of the Literature. Qual Health Res. 2020 Aug;30(10):1596-1604. doi: 10.1177/1049732320921835. PMID 32667277
- [Background] Umaña-Taylor AJ, Yazedjian A, Bámaca-Gómez MY. Developing the Ethnic Identity Scale using Eriksonian and social identity perspectives. Identity Int J Theory Res. 2004;4:9-38.
- [Background] Berkel C, Knight GP, Zeiders KH, Tein JY, Roosa MW, Gonzales NA, Saenz D. Discrimination and adjustment for Mexican American adolescents: A prospective examination of the benefits of culturally-related values. J Res Adolesc. 2010 Nov 15;20(4):893-915. doi: 10.1111/j.1532-7795.2010.00668.x. PMID 21359093
- [Background] Kulish AL, Cavanaugh AM, Stein GL, Kiang L, Gonzalez LM, Supple A, Mejia Y. Ethnic-racial socialization in Latino families: The influence of mothers' socialization practices on adolescent private regard, familism, and perceived ethnic-racial discrimination. Cultur Divers Ethnic Minor Psychol. 2019 Apr;25(2):199-209. doi: 10.1037/cdp0000222. Epub 2018 Oct 4. PMID 30284851
- [Background] Yasui M, Dishion TJ. Direct observation of family management: validity and reliability as a function of coder ethnicity and training. Behav Ther. 2008 Dec;39(4):336-47. doi: 10.1016/j.beth.2007.10.001. Epub 2008 Apr 20. PMID 19027430
- [Background] Achenbach TM. Manual for the Youth Self-Report and 1991 Profile. Department of Psychiatry, University of Vermont;1991
- [Background] Achenbach TM, Edelbrock C. Child behavior checklist. Burlington. 1991;7:371-392.
- [Background] Irwin DE, Gross HE, Stucky BD, Thissen D, DeWitt EM, Lai JS, Amtmann D, Khastou L, Varni JW, DeWalt DA. Development of six PROMIS pediatrics proxy-report item banks. Health Qual Life Outcomes. 2012 Feb 22;10:22. doi: 10.1186/1477-7525-10-22. PMID 22357192
- [Background] Irwin DE, Stucky B, Langer MM, Thissen D, Dewitt EM, Lai JS, Varni JW, Yeatts K, DeWalt DA. An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Qual Life Res. 2010 May;19(4):595-607. doi: 10.1007/s11136-010-9619-3. Epub 2010 Mar 7. PMID 20213516
- [Background] McDermott ER, Umaña-Taylor AJ, Martinez-Fuentes S. Measuring Latino adolescents' coping with ethnic-racial discrimination. J Psychoeduc Assess. 2019;37(6):730-742.
- [Background] Hughes D, Chen L. When and what parents tell children about race: An examination of race-related socialization among African American families. Appl Dev Sci. 1997;1(4):200-214. doi:10.1207/S1532480XADS0104_4
- [Background] Christophe NK, Stein GL, Kiang L. A 21st Century take on patterns of racial-ethnic socialization: Competency and content among minoritized parents. Soc Sci. 2022;11(2).
- [Background] Jones SCT, Christophe NK, Stevenson HC, Stein GL, Kiang L, Chan M, Anderson RE. We got this: Evaluating racial socialization competency among diverse ethnic-racial groups. J Fam Psychol. 2024 Jun;38(4):571-581. doi: 10.1037/fam0001210. Epub 2024 Apr 4. PMID 38573697
- [Background] Anderson RE, Jones SCT, Stevenson HC. The initial development and validation of the Racial Socialization Competency Scale: Quality and quantity. Cultur Divers Ethnic Minor Psychol. 2020 Oct;26(4):426-436. doi: 10.1037/cdp0000316. Epub 2019 Dec 30. PMID 31886685
- [Background] Miller WR, Johnson WR. A natural language screening measure for motivation to change. Addict Behav. 2008 Sep;33(9):1177-82. doi: 10.1016/j.addbeh.2008.04.018. Epub 2008 May 9. PMID 18558466
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Li AE, Jhawar S, Grignol V, Agnese D, Oppong BA, Beyer S, Bazan JG, Skoracki R, Shen C, Park KU. Implementation of a Breast Intraoperative Oncoplastic Form to Aid Management of Oncoplastic Surgery. J Surg Res. 2023 Oct;290:9-15. doi: 10.1016/j.jss.2023.04.002. Epub 2023 May 8. PMID 37163831
- [Background] Birk JL, Cumella R, Lopez-Veneros D, Agarwal S, Kronish IM. Feasibility of a remote heart rate variability biofeedback intervention for reducing anxiety in cardiac arrest survivors: A pilot trial. Contemp Clin Trials Commun. 2024 Jan 8;37:101251. doi: 10.1016/j.conctc.2023.101251. eCollection 2024 Feb. PMID 38312473
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Dishion TJ, Hogansen J, Winter C, Jabson J. The Coder Impressions Inventory. In Child and Family Center, University of Oregon; 2004.
- [Background] Douglass S, Umana-Taylor AJ. Time-varying effects of family ethnic socialization on ethnic-racial identity development among Latino adolescents. Dev Psychol. 2016 Nov;52(11):1904-1912. doi: 10.1037/dev0000141. Epub 2016 Oct 6. PMID 27709995
- [Background] Umaña-Taylor AJ, Hill NE. Ethnic-racial socialization in the family: A decade's advance on precursors and outcomes. J Marriage Fam. 2020;82(1):244-271.
- [Background] Baldwin-White AJM, Kiehne E, Umana-Taylor A, Marsiglia FF. In Pursuit of Belonging: Acculturation, Perceived Discrimination, and Ethnic-Racial Identity among Latino Youths. Soc Work Res. 2017 Mar;41(1):43-52. doi: 10.1093/swr/svw029. Epub 2017 Jan 10. PMID 28533677
- [Background] Leary M, Cacchione PZ, Demiris G, Carthon JMB, Bauermeister JA. An integrative review of human-centered design and design thinking for the creation of health interventions. Nurs Forum. 2022 Nov;57(6):1137-1152. doi: 10.1111/nuf.12805. Epub 2022 Oct 18. PMID 36255150
- [Background] Lyon AR, Brewer SK, Arean PA. Leveraging human-centered design to implement modern psychological science: Return on an early investment. Am Psychol. 2020 Nov;75(8):1067-1079. doi: 10.1037/amp0000652. PMID 33252945
- [Background] Dishion TJ, Shaw D, Connell A, Gardner F, Weaver C, Wilson M. The family check-up with high-risk indigent families: preventing problem behavior by increasing parents' positive behavior support in early childhood. Child Dev. 2008 Sep-Oct;79(5):1395-414. doi: 10.1111/j.1467-8624.2008.01195.x. PMID 18826532
- [Background] Shaw DS, Galan CA, Lemery-Chalfant K, Dishion TJ, Elam KK, Wilson MN, Gardner F. Trajectories and Predictors of Children's Early-Starting Conduct Problems: Child, Family, Genetic, and Intervention Effects. Dev Psychopathol. 2019 Dec;31(5):1911-1921. doi: 10.1017/S0954579419000828. PMID 31370912
- [Background] Aguayo L, Hernandez IG, Yasui M, Estabrook R, Anderson EL, Davis MM, Briggs-Gowan MJ, Wakschlag LS, Heard-Garris N. Cultural socialization in childhood: Analysis of parent-child conversations with a direct observation measure. J Fam Psychol. 2021 Mar;35(2):138-148. doi: 10.1037/fam0000663. PMID 33871275
- [Background] Yasui M. Observed ethnic-racial socialization and early adolescent adjustment. University of Oregon; 2008.
- [Background] Dishion TJ, Nelson SE, Kavanagh K. The family check-up with high-risk young adolescents: Preventing early-onset substance use by parent monitoring. Behav Ther. 2003;34(4):553-571. doi:10.1016/S0005- 7894(03)80035-7
- [Background] Anderson RE, McKenny MC, Stevenson HC. EMBRace: Developing a Racial Socialization Intervention to Reduce Racial Stress and Enhance Racial Coping among Black Parents and Adolescents. Fam Process. 2019 Mar;58(1):53-67. doi: 10.1111/famp.12412. Epub 2018 Dec 15. PMID 30552778
- [Background] Smalls C. Effects of mothers' racial socialization and relationship quality on African American youth's school engagement: a profile approach. Cultur Divers Ethnic Minor Psychol. 2010 Oct;16(4):476-84. doi: 10.1037/a0020653. PMID 21058810
- [Background] Frabutt JM, Walker AM, MacKinnon-Lewis C. Racial Socialization Messages and the Quality of Mother/Child Interactions in African American Families. J Early Adolesc. 2002;22(2):200-217. doi:10.1177/0272431602022002004
- [Background] Smith-Bynum MA, Anderson RE, Davis BL, Franco MG, English D. Observed Racial Socialization and Maternal Positive Emotions in African American Mother-Adolescent Discussions About Racial Discrimination. Child Dev. 2016 Nov;87(6):1926-1939. doi: 10.1111/cdev.12562. Epub 2016 May 23. PMID 27211821
- [Background] Yasui M. A review of the empirical assessment of processes in ethnic-racial socialization: Examining methodological advances and future areas of development. Dev Rev. 2015;37:1-40. doi:10.1016/j.dr.2015.03.001
- [Background] Schunk DH. Goal setting and self-efficacy during self-regulated learning. Educ Psychol. 1990;25(1):71- 86.
- [Background] Zimmerman BJ. A social cognitive view of self-regulated academic learning. J Educ Psychol. 1989;81(3):329-339.
- [Background] Bandura A. Social-learning theory of identificatory processes. Handb Social Theory Res. 1969;213.
- [Background] Bakermans-Kranenburg MJ, van IJzendoorn MH, Juffer F. Less is more: meta-analyses of sensitivity and attachment interventions in early childhood. Psychol Bull. 2003 Mar;129(2):195-215. doi: 10.1037/0033-2909.129.2.195. PMID 12696839
- [Background] Galan CA, Shaw DS, O'Rourke F, Reynolds MD, Gill A, Bogen DL, Ridenour TA. Substance Use Screening and Prevention for Adolescents in Pediatric Primary Care: A Randomized Clinical Trial using the Family Check-Up. Res Child Adolesc Psychopathol. 2023 Feb;51(2):151-163. doi: 10.1007/s10802-022-00978-2. Epub 2022 Oct 8. PMID 36208361
- [Background] Yagmur S, Mesman J, Malda M, Bakermans-Kranenburg MJ, Ekmekci H. Video-feedback intervention increases sensitive parenting in ethnic minority mothers: a randomized control trial. Attach Hum Dev. 2014;16(4):371-86. doi: 10.1080/14616734.2014.912489. PMID 24972105
- [Background] Balldin S, Fisher PA, Wirthberg I. Video feedback intervention with children: A systematic review. Res Soc Work Pract. 2016;28(6):682-695.
- [Background] Neblett Jr. EW, White RL, Ford KR, Philip CL, Nguyên HX, Sellers RM. Patterns of racial socialization and psychological adjustment: Can parental communications about race reduce the impact of racial discrimination? J Res Adolesc. 2008;18(3):477-515.
- [Background] Telzer EH. Skin color and self-perceptions of immigrant and U.S.-born Latinas. Hisp J Behav Sci. 2009;31(3):357-374.
- [Background] Hughes D, Rodriguez J, Smith EP, Johnson DJ, Stevenson HC, Spicer P. Parents' ethnic-racial socialization practices: a review of research and directions for future study. Dev Psychol. 2006 Sep;42(5):747-70. doi: 10.1037/0012-1649.42.5.747. PMID 16953684
- [Background] Priest N, Walton J, White F, Kowal E, Baker A, Paradies Y. Understanding the complexities of ethnicracial socialization processes for both minority and majority groups: A 30-year systematic review. Int J Intercult Relat. 2014;43:139-155. doi:10.1016/j.ijintrel.2014.08.003
- [Background] Gonzalez LM, Martin Romero MY, Stein GL, Coard SI, Kiang L. Troubled waters: Barriers to preparation for bias conversations across racially/ethnically diverse families. Fam Relat. Published online 2022.
- [Background] González AG, Umaña-Taylor AJ, Bámaca MY. Familial ethnic socialization among adolescents of Latino and European descent: Do Latina mothers exert the most influence? J Fam Issues. 2006;Feb;27(2):184-207.
- [Background] Zeiders KH, Umana-Taylor AJ, Martinez-Fuentes S, Updegraff KA, Bayless SD, Jahromi LB. Latina/o Youths' Discrimination Experiences in the U.S. Southwest: Estimates from Three Studies. Appl Dev Sci. 2021;25(1):51-61. doi: 10.1080/10888691.2018.1527695. Epub 2018 Dec 20. PMID 33716491
- [Background] Hernandez MM, Conger RD, Robins RW, Bacher KB, Widaman KF. Cultural socialization and ethnic pride among Mexican-origin adolescents during the transition to middle school. Child Dev. 2014 Mar-Apr;85(2):695-708. doi: 10.1111/cdev.12167. Epub 2013 Sep 30. PMID 24117445
- [Background] Huynh VW, Fuligni AJ. Ethnic socialization and the academic adjustment of adolescents from Mexican, Chinese, and European backgrounds. Dev Psychol. 2008 Jul;44(4):1202-8. doi: 10.1037/0012-1649.44.4.1202. PMID 18605847
- [Background] Hughes D, Hagelskamp C, Way N, Foust MD. The role of mothers' and adolescents' perceptions of ethnic-racial socialization in shaping ethnic-racial identity among early adolescent boys and girls. J Youth Adolesc. 2009 May;38(5):605-26. doi: 10.1007/s10964-009-9399-7. Epub 2009 Mar 17. PMID 19636759
- [Background] Araujo Dawson B, Quiros L. The effects of racial socialization on the racial and ethnic identity development of Latinas. J Lat Psychol. 2014;2(4):200-213. doi:10.1037/lat0000024
- [Background] Gonzalez LM, Stein GL, Martin-Romero MY, Coard SI, Kiang L. Why we don't talk about it: A crosscultural exploration of the barriers to prep for bias conversations among families from minoritized racial/ethnic groups. In: Society for Research in Child Development (SRCD); 2020.
- [Background] Priest N, Paradies Y, Trenerry B, Truong M, Karlsen S, Kelly Y. A systematic review of studies examining the relationship between reported racism and health and wellbeing for children and young people. Soc Sci Med. 2013 Oct;95:115-27. doi: 10.1016/j.socscimed.2012.11.031. Epub 2012 Dec 19. PMID 23312306
- [Background] Anderson RE, Stevenson HC. RECASTing racial stress and trauma: Theorizing the healing potential of racial socialization in families. Am Psychol. 2019 Jan;74(1):63-75. doi: 10.1037/amp0000392. PMID 30652900
- [Background] McDermott ER, Umana-Taylor AJ, Zeiders KH. Profiles of Coping with Ethnic-Racial Discrimination and Latina/o Adolescents' Adjustment. J Youth Adolesc. 2019 May;48(5):908-923. doi: 10.1007/s10964-018-0958-7. Epub 2018 Nov 23. PMID 30471057
- [Background] Fernandez ME, Ruiter RAC, Markham CM, Kok G. Intervention Mapping: Theory- and Evidence-Based Health Promotion Program Planning: Perspective and Examples. Front Public Health. 2019 Aug 14;7:209. doi: 10.3389/fpubh.2019.00209. eCollection 2019. PMID 31475126
- [Background] Fukkink RG. Video feedback in widescreen: a meta-analysis of family programs. Clin Psychol Rev. 2008 Jul;28(6):904-16. doi: 10.1016/j.cpr.2008.01.003. Epub 2008 Feb 5. PMID 18359136
- [Background] Coard SI, Wiley KC, Evans AG. The Black Parenting Strengths and Strategies Program-Racialized Short (BPSS-RS): "Real-world" dismantle, implementation, and evaluation. Advers Resil Sci. 2021;2(4):235-245.
- [Background] Coard SI, Herring MH, Watkins MH, Foy-Watson SA, McCoy SZ. Black Parents Strengths and Strategies (BPSS) program: A cultural adaptation of the strong-willed child program. In: Handbook of Culturally Responsive School Mental Health. Springer; 2013.
- [Background] Anderson RE, Jones SCT, Navarro CC, McKenny MC, Mehta TJ, Stevenson HC. Addressing the Mental Health Needs of Black American Youth and Families: A Case Study from the EMBRace Intervention. Int J Environ Res Public Health. 2018 May 2;15(5):898. doi: 10.3390/ijerph15050898. PMID 29724068
- [Background] Brody GH, Murry VM, Gerrard M, Gibbons FX, Molgaard V, McNair L, Brown AC, Wills TA, Spoth RL, Luo Z, Chen YF, Neubaum-Carlan E. The Strong African American Families Program: translating research into prevention programming. Child Dev. 2004 May-Jun;75(3):900-17. doi: 10.1111/j.1467-8624.2004.00713.x. PMID 15144493
- [Background] Stein GL, Coard SI, Gonzalez LM, Kiang L, Sircar JK. One talk at a time: Developing an ethnic-racial socialization intervention for Black, Latinx, and Asian American families. J Soc Issues. 2021;77(4):1014-1036.
- [Background] Huguley JP, Wang MT, Vasquez AC, Guo J. Parental ethnic-racial socialization practices and the construction of children of color's ethnic-racial identity: A research synthesis and meta-analysis. Psychol Bull. 2019 May;145(5):437-458. doi: 10.1037/bul0000187. Epub 2019 Mar 21. PMID 30896188
- [Background] Wang MT, Henry DA, Smith LV, Huguley JP, Guo J. Parental ethnic-racial socialization practices and children of color's psychosocial and behavioral adjustment: A systematic review and meta-analysis. Am Psychol. 2020 Jan;75(1):1-22. doi: 10.1037/amp0000464. Epub 2019 May 6. PMID 31058521
- [Background] Ayón C, Nieri T, Ruano E. Ethnic-racial socialization among Latinx families: A systematic review of the literature. Soc Serv Rev. 2020;94(4):693-747.
- [Background] Trent M, Dooley DG, Douge J; SECTION ON ADOLESCENT HEALTH; COUNCIL ON COMMUNITY PEDIATRICS; COMMITTEE ON ADOLESCENCE. The Impact of Racism on Child and Adolescent Health. Pediatrics. 2019 Aug;144(2):e20191765. doi: 10.1542/peds.2019-1765. PMID 31358665
- [Background] Benner AD, Wang Y, Shen Y, Boyle AE, Polk R, Cheng YP. Racial/ethnic discrimination and well-being during adolescence: A meta-analytic review. Am Psychol. 2018 Oct;73(7):855-883. doi: 10.1037/amp0000204. Epub 2018 Jul 19. PMID 30024216
- [Background] Greene ML, Way N, Pahl K. Trajectories of perceived adult and peer discrimination among Black, Latino, and Asian American adolescents: patterns and psychological correlates. Dev Psychol. 2006 Mar;42(2):218-36. doi: 10.1037/0012-1649.42.2.218. PMID 16569162
- [Background] Stein GL, Castro-Schilo L, Cavanaugh AM, Mejia Y, Christophe NK, Robins R. When Discrimination Hurts: The Longitudinal Impact of Increases in Peer Discrimination on Anxiety and Depressive Symptoms in Mexican-origin Youth. J Youth Adolesc. 2019 May;48(5):864-875. doi: 10.1007/s10964-019-01012-3. Epub 2019 Mar 16. PMID 30879164
- [Background] Edwards LM, Romero AJ. Coping with discrimination among Mexican descent adolescents. Hisp J Behav Sci. 2008;30(1):24-39.
- [Background] Flores E, Tschann JM, Dimas JM, Pasch LA, de Groat CL. Perceived racial/ethnic discrimination, posttraumatic stress symptoms, and health risk behaviors among Mexican American adolescents. J Couns Psychol. 2010 Jul;57(3):264-73. doi: 10.1037/a0020026. PMID 21133578

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT07055906/Prot_SAP_000.pdf